CLINICAL TRIAL: NCT03168126
Title: Advanced Hemodynamic Monitoring in Free Flap Surgery
Acronym: AHM
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: 002
Record Dates: First submitted 2017-05-24; First posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Hemodynamic Rebound; Volume Overload; Fluid Overload; Bloodpressure
MeSH Terms: conditions — Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pro-AQT-Monitoting: Patients with OSCC of the jaws and tumor resection + primary free flap reconstruction
  Interventions: Device: Pro-AQT

INTERVENTIONS:
Device: Pro-AQT — Use of the device for advanced hemodynamic monitoring

SUMMARY:
Background: Anesthesia in free flap surgery is challenging. Monitoring of hemodynamic changes and their influence on the cardiovascular system in permanent feedback loops allow control, which is what anesthesiologists aim for to ensure an adequate blood flow and tissue oxygenation. The circulatory support and inferable volume administration are managed via heart rate (HR) and mean arterial pressure (MAP), but both parameters are influenced by variable components and are thus unfavorable for volume management. The aim of this study was to evaluate whether volume requirement may be assumable to additional monitoring parameters.

Methods: 31 patients were enrolled prospectively. HR, MAP, central venous pressure and O2 saturation were comprehended based on the protocols. We expanded the data set by a permanent blinded intraoperative monitoring with registration of the Cardiac Index (CI) and Stroke Volume Variation (SVV) and semi-invasive pulse-contour analysis utilizing the Pro-AQT-Device.

DETAILED DESCRIPTION:
We conducted a prospective cohort study in accordance with the WMA Declaration of Helsinki. Standard general anesthesia with intubation and administration of sufentanil, propofol and esmeron relaxant was performed in all patients undergoing primary free flap reconstruction in course of a head and neck tumor reconstruction. Hemodynamic monitoring measurement of cardiac index and the parameter stroke volume variation as surrogate for cardiac pre-load was performed using a Pro-AQT Monitor. Using an arterial catheter previously set by the Seldinger technique as part of the standard equipment, the mean, diastolic and systolic arterial pressure was measured as part of the standard monitoring as presented. This tube was previously deaerated and flushed with 2% NaCl and connected in series with a sensor, which passes over electric line signals to the Pro-AQT-Monitor®. Based on previously entered patient data and an analysis of the arterial pulse curve characteristics, a cardiac index (CI) start-value is determined by the system. The sampling of the arterial pressure characteristics is affected by a signal having a frequency of 250 Hz. The start value is the basis for the further determination of HI trend values. The arterial pulse contour is continuously tapped and analyzed and offset against the determined start value. To calculate the cardiac index, the PICCO®-pulse contour algorithm is applied. Every 12 seconds, a new measurement is performed and documented by the system.

From the read logs ProAQT Monitor® the values of the CI, MAP, HR, stroke volume index (SVI), the stroke volume variation (SVV) and the systemic resistance index (SRI) were recorded at different measurement intervals throughout the operation. All parameters were evaluated for volume control in the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age, free flap surgery, oral squamous cell carcinoma, informed consent

Exclusion Criteria:

* <18 years of age, no informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with oral squamous cell carcinoma undergoing tumor resection + primary reconstruction with a free flap
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Stroke Volume Variance (SVV) | during the surgical intervention

SECONDARY OUTCOMES:
Mean arterial pressure | during the surgical intervention
heart rate | during the surgical intervention
cardiac index | during the surgical intervention
standard resistance index | during the surgical intervention

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Wikner, MD DMD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wakeling HG, McFall MR, Jenkins CS, Woods WG, Miles WF, Barclay GR, Fleming SC. Intraoperative oesophageal Doppler guided fluid management shortens postoperative hospital stay after major bowel surgery. Br J Anaesth. 2005 Nov;95(5):634-42. doi: 10.1093/bja/aei223. Epub 2005 Sep 9. PMID 16155038